CLINICAL TRIAL: NCT05857332
Title: A Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SG1906 in Patients With CLDN18.2-Positive Locally Advanced Unresectable or Metastatic Solid Tumors.
Brief Title: SG1906 for CLDN18.2-Positive Solid Tumors
Acronym: CSG-1906-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSG-1906-101
Record Dates: First submitted 2023-04-23; First posted 2023-05-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Unresectable or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SG1906 (Experimental): SG1906 monotherapy intravenous (IV) infusion - Biweekly doses
  Interventions: Drug: SG1906

INTERVENTIONS:
Drug: SG1906 — Phase 1a will use an accelerated titration-Bayesian optimal interval (AT-BOIN) design with 7 dose cohorts: 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 6 mg/kg, 9 mg/kg, and 12 mg/kg by IV infusion. Accelerated titration (i.e., 1 patient each) will be applied to the first 2 cohorts.

SUMMARY:
This is a Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SG1906 in Patients with CLDN18.2-Positive Locally Advanced Unresectable or Metastatic Solid Tumors.

DETAILED DESCRIPTION:
After a screening period of up to 28 days for each study phase, qualified patients will be enrolled to receive their assigned dose of SG1906, administered every 2 weeks (Q2W), until disease progression or intolerable toxicity, starting of a new anticancer treatment, withdrawal of consent, lost to follow up, death, or end of the study, whichever occurs first.

Phase Ia: Dose-escalation Stage The study population in Phase Ia includes patients with CLDN18.2-positive histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumor who have relapsed after standard therapy, have failed standard therapy, are intolerant to standard therapy, are not eligible for standard therapy, or refuse standard therapy. Phase Ib: Dose-expansion Stage The study population in this phase will include patients with histologically or cytologically confirmed CLDN18.2-positive locally advanced unresectable or metastatic G/GEJ cancer or PC who have failed to respond to standard therapy, have relapsed after standard therapy, or are intolerant to standard therapy; and who have disease progression as confirmed by the Investigator or documented by medical history.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following criteria to be eligible for participation in this study:

  1. Understand and voluntarily sign the informed consent form (ICF).
  2. Age ≥18 years.
  3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
  4. Expected survival time of ≥3 months.
  5. Able to provide tumor tissue samples for CLDN18.2 detection.
  6. Specific requirements for patients enrolled in Phase Ia and Phase Ib are as follows:

     Phase Ia Dose Escalation Phase
     1. Patients with CLDN18.2-positive histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumor who have relapsed after standard therapy, have failed standard therapy, are intolerant to standard therapy, are not eligible for standard therapy, or refuse standard therapy.
     2. CLDN18.2 positivity is defined as H score ≥1 by central laboratory immunohistochemistry.

     Phase Ib Dose Expansion Stage
     1. Patients with histologically or cytologically confirmed CLDN18.2-positive locally advanced unresectable or metastatic G/GEJ adenocarcinoma or pancreatic cancer who have failed to respond to standard therapy, have relapsed after standard therapy, or are intolerant to standard therapy.
     2. CLDN18.2 positivity is defined as H score ≥40 by central laboratory immunohistochemistry.
  7. At least one evaluable lesion (refer to Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1]).
  8. Adequate function of vital organs, defined as follows:

     1. Bone marrow function (no transfusion, erythropoietin, granulocyte colony-stimulating factor, or other medically supportive therapy within 7 days prior to the first dose): neutrophil count ≥1.5 × 109/L, platelet count ≥100 × 109/L, and hemoglobin level ≥10.0 g/dL.
     2. Adequate liver function, which must meet all of the following criteria:

        * Serum total bilirubin ≤1.5 × upper limit of normal (ULN).
        * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (AST and ALT ≤5 × ULN in patients with liver metastases).
        * Albumin ≥3.0 g/L.
     3. Renal function: serum creatinine ≤1.5 × ULN or endogenous creatinine clearance ≥50 mL/min (Cockcroft-Gault formula).
     4. Coagulation: international normalized ratio ≤1.5 × ULN or prothrombin time ≤1.5 × ULN, activated partial thromboplastin time ≤1.5 × ULN without receiving anticoagulation therapy.
  9. Toxicity caused by prior anti-tumor therapy recovered to Grade 0 to 1 (CTCAE 5.0), except for alopecia, Grade ≤2 sensory neuropathy, lymphocytopenia, and endocrine disorders controlled with hormone replacement therapy.
  10. Female patients of childbearing potential and male patients whose female partners are of childbearing potential need to use at least one approved contraceptive (e.g., intrauterine device, pill, or condom) during study treatment and for at least 6 months (180 days) after the last dose; female patients of childbearing potential must have a negative blood human chorionic gonadotropin (HCG) test within 7 days prior to dosing and must not be lactating.
  11. Male patients must refrain from donating sperm from the time the ICF is signed until at least 6 months after the last dose.

Exclusion Criteria:

Patients who meet any of the following criteria cannot be enrolled:

1. Presence of active central nervous system metastatic lesions; presence of metastases to the brainstem or meninges, spinal cord metastases or compression. Exception: patients with previously treated brain metastases (e.g., surgery, radiation therapy) who are clinically stable for at least 4 weeks after treatment (calculated from the first dose of investigational drug) and have discontinued corticosteroids for ≥14 days prior to the administration of investigational drug; patients with untreated, asymptomatic brain metastases (i.e., no neurological symptoms, no need for corticosteroids, brain metastases ≤1.5 cm in length, no significant edema around the brain metastases).
2. Active autoimmune disease requiring systemic therapy within the past 2 years (e.g., use of immunomodulatory drugs, corticosteroids, or immunosuppressive medications); related replacement therapy is allowed (e.g., thyroid hormone, insulin, or physiologic corticosteroid replacement for renal or pituitary insufficiency).
3. Pyloric obstruction or any other condition that can cause long-term chronic nausea, persistent recurrent vomiting (≥3 vomit episodes in 24 hours) or diarrhea.
4. Patients who have recently developed gastrointestinal bleeding (i.e., a history of hematemesis, hematochezia, or melena within the past 3 months) without evidence of recovery confirmed by endoscopy or colonoscopy; or patients with evidence of risk of gastric bleeding.
5. Patients with active gastrointestinal disease including, but not limited to, gastric or duodenal ulcers, acute gastric or intestinal perforation, acute necrotizing pancreatitis, ulcerative enteritis, congenital megacolon or Crohn's disease.
6. Patients requiring long-term treatment with non-steroidal anti-inflammatory drugs (NSAIDs); patients who are using anticoagulants such as heparin at therapeutic doses or vitamin K antagonists (except for prophylaxis).
7. Presence of body fluid (hydrothorax, ascites, pericardial effusion, etc.) requiring local treatment or repeated drainage.
8. Unintentional weight loss ≥5% within 1 month prior to initial dose, even with peripheral or central intravenous nutritional support.
9. History of hemolytic anemia from any cause (including Evans syndrome).
10. History of defects in red blood cell production, hemoglobin production, or metabolism, such as glucose-6-phosphate dehydrogenase deficiency, thalassemia, sickle cell disease, and hereditary spherocytosis.
11. History of hemophagocytic lymphohistiocytosis.
12. Presence of active infection requiring antibiotic therapy within 2 weeks prior to the first dose, except for prophylaxis.
13. Presence of cardiovascular system disease within 6 months prior to screening that meets any of the following:

    1. Cardiac function: congestive heart failure of New York Heart Association (NYHA) class III or IV; left ventricular ejection fraction <50%.
    2. Clinically significant cardiac disease or surgery within 6 months prior to the first dose of the investigational drug, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, coronary/peripheral artery bypass, etc.
    3. QTcF (corrected QT interval with Fridericia formula) >450 ms in men and >470 ms in women; history of clinically significant ventricular arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, tip-twist ventricular tachycardia); history or family history of congenital long QT syndrome; arrhythmias requiring antiarrhythmic drug therapy (patients with atrial fibrillation with controllable heart rate 1 month prior to the first dose of the investigational drug may be enrolled).
    4. History of arterial thrombosis, deep venous thrombosis and pulmonary embolism within 6 months prior to the first dose.
14. Hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg) that has not been effectively controlled after treatment with standardized antihypertensive medication.
15. Patients with active hepatitis B or C. In case of positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (HBcAb) during the screening period, further hepatitis B virus (HBV) DNA titer testing must be performed (HBV DNA≤200 IU/mL is required). Patients who are positive for hepatitis C virus (HCV) must receive further HCV RNA testing (no higher than the upper limit of the detection value at their study site); patients may be enrolled in the study only after active hepatitis B or C requiring treatment has been excluded.
16. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV antibody positive);
17. Known history of Grade 3 to 4 hypersensitivity reactions to any biological product, history of life threatening hypersensitivity reactions, or known hypersensitivity to components of SG1906 drug product (Grade ≥3 hypersensitivity reactions).
18. Have received any of the following treatments or procedures:

    1. Prior treatment with any antitumor therapy targeting CLDN18.2 or CD47
    2. Patients who have undergone open surgery ≤3 months prior to the first dose (except for surgeries for the purpose of biopsy).
    3. Prior allogeneic organ grafting.
    4. Systemic anticancer therapy (including chemotherapy, targeted therapy, hormonal therapy and immunotherapy) within 28 days or 5 drug half-lives (whichever is shorter) prior to the first dose of the investigational drug, and all AEs have not returned to grade ≤1 (CTCAE 5.0), except for alopecia.
    5. Radiotherapy ≤14 days prior to the first dose of the investigational drug; palliative radiotherapy is allowed if it is completed within 2 weeks prior to the enrollment in the study and radiotherapy-related toxicity has recovered to grade ≤1 (CTCAE 5.0), except for alopecia
    6. Any live vaccine within 4 weeks prior to the first dose of the investigational drug
    7. Have received treatment with various growth factors, blood transfusions or other blood products for anemia or decreased platelet count within 14 days prior to the first dose of the investigational drug.
19. Have received systemic corticosteroids (at a dose equivalent to >10 mg/day prednisone) or other immunosuppressive drugs within 14 days prior to the first dose. The following are permitted:

    1. Topical or inhaled glucocorticoids in physiologic replacement doses are allowed
    2. The use of short-course (≤7 days) corticosteroids at physiologic replacement doses for the prevention or treatment of non-autoimmune diseases is allowed.
20. Any other condition that, in the opinion of the Investigator, may lead to inappropriate participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of one year
  Number and percentage of AE which is calculated by worst CTCAE grade by CTCAE 5.0
MTD/MAD/ RP2D | Through study completion, an average of one year
  To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) for intravenous (IV) administration of SG1906 in patients with CLDN18.2-positive locally advanced unresectable or metastatic solid tumors.; To preliminarily determine the recommended Phase 2 dose (RP2D) of SG1906 given intravenously in patients with CLDN18.2-positive locally advanced unresectable or metastatic solid tumors.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): AUC | Through study completion, an average of one year
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Pharmacokinetics (PK): Cmax | Through study completion, an average of one year
  Cmax to maximum drug concentration.
Pharmacokinetics (PK):limination half-life (T1/2) | Through study completion, an average of one year
  limination half-life (T1/2) of the drug after administration.
receptor occupancy (RO) | Through study completion, an average of one year
  receptor occupancy (RO) of CD47 on the surface of peripheral blood cells;
Immunogenicity endpoints: | Through study completion, an average of one year
  levels of anti-drug antibodies (ADAs) and neutralizing antibodies (tested in ADA-positive samples only).
Efficacy endpoints: | Through study completion, an average of one year
  objective response rate (ORR).

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Xiamen University, Xiamen, Fujian
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No